CLINICAL TRIAL: NCT06288165
Title: Coronary Sinus Reducer Implantation for Refractory Angina - Long-Term Evaluation of Device Safety and Efficacy- Lower Silesia Sinus Reducer Registry (LSSRR)
Brief Title: Lower Silesia Sinus Reducer Registry
Acronym: LSSRR
Status: Recruiting | Type: Observational
Sponsor: Regional Cardiology Center, The Copper Health Centre (MCZ), (Other)
Responsible Party: Principal Investigator, Adrian Włodarczak, Profesaor, Regional Cardiology Center, The Copper Health Centre (MCZ),
Other Study IDs: CopperHealthCentre2
Record Dates: First submitted 2024-02-18; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Safety Issues; Efficacy, Self
Keywords: Coronary Sinus Reducer; Refractory angina; Chronic coronary artery diseases (CAD); Non-obstructive Coronary artery diseases (CAD); Coronary microvascular dysfunction
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Coronary Sinus Reducer implantation: Subject after Coronary Sinus Reducer implantation due to chronic disabling refractory angina pectoris (Canadian Cardiovascular Society [CCS] classes 2-4) despite maximally tolerated anti-angina medical therapy. All patients were evaluated by the local Heart Team and considered not amenable to percutaneous or surgical revascularization procedures. After the Heart Team evaluation patients were qualified for the procedure or Coronary Sinus Reducer implantation unless they meet one of the exclusion criteria. Initial patient evaluation (prior to device implantation) consists of past medical history, actual clinical assessment with an evaluation of CCS class, Seattle Angina Questionnaire - 7 items (SAQ-7) scores, 6-min walk distance (6-MWT) test, and echocardiography. First, a follow-up visit is scheduled 1 month after the implantation procedure than the follow-up is planned twice a year.
  Interventions: Device: Coronary Sinus Reducer Implantation

INTERVENTIONS:
Device: Coronary Sinus Reducer Implantation — Coronary Sinus (CS) Reducer implantation to coronary sinus via the venous system. Coronary Sinus is a balloon-expandable, hourglass-shaped, scaffold implanted percutaneously into the coronary sinus creating a narrowing to delay blood outflow.

SUMMARY:
Lower Silesia Sinus Reducer Registry is a , single-center, single-arm registry including patients with chronic disabling refractory angina pectoris (Canadian Cardiovascular Society [CCS] classes 2-4) despite maximally tolerated anti-angina medical therapy who underwent Coronary Sinus Reducer implantation .

DETAILED DESCRIPTION:
Lower Silesia Sinus Reducer Registry is a single-center, single-arm registry including all consecutive patients who were referred to the Cardiac Department of Copper Health Center due to chronic disabling refractory angina pectoris (Canadian Cardiovascular Society [CCS] classes 2-4) despite maximally tolerated anti-angina medical therapy and underwent Coronary Sinus Reducer implantation. All patients were evaluated by the local Heart Team and considered not amenable to percutaneous or surgical revascularization procedures. After the Heart Team evaluation patients were qualified for the procedure or Coronary Sinus Reducer implantation unless they met one of the exclusion criteria.

Initial patient evaluation (prior to device implantation) consisted of past medical history, actual clinical assessment with an evaluation of CCS class, Seattle Angina Questionnaire - 7 items (SAQ-7) scores, 6-min walk distance (6-MWT) test, and echocardiography. First, a follow-up visit was scheduled 1 month after the implantation procedure.The study will include clinical assessments every six months during an observation period. The primary outcomes will be gathered one year after the implantation of the CS. Nevertheless, clinical follow-up will continue for up to five years after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. present of chronic disabling refractory angina pectoris (Canadian Cardiovascular Society [CCS] classes 2-4) despite maximally tolerated anti-angina medical therapy
2. Heart team evaluation with consideration of ineligibility for percutaneous or surgical revascularization procedures.

Exclusion Criteria:

1. recent acute coronary syndrome (<3 months),
2. recent coronary revascularization (<3 months)
3. a mean right atrial pressure higher than 15 mm Hg
4. coronary sinus proximal diameter <10mm and >14mm
5. life expectancy under 12 months,
6. advanced heart failure (New York Heart Association [NYHA] Classification - classes 3-4),
7. potential implantable cardiac resynchronization therapy defibrillator (CRT-D) implantation candidate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of subjects with chronic disabling refractory angina pectoris (Canadian Cardiovascular Society [CCS] classes 2-4) who have not responded to treatment with maximally tolerated anti-angina medical therapy. The local Heart Team will evaluate all patients and determine that they are not suitable for percutaneous or surgical revascularization procedures. Following the Heart Team evaluation, patients who do not have any revascularization options available to them are eligible for the procedure or Coronary Sinus Reducer implantation, unless they meet one of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2027-05-11 (Estimated); Study Completion 2027-05-11 (Estimated)

PRIMARY OUTCOMES:
The Clinical success - reduction of angina symptoms | 1-Year after implantation
  The severity of angina is assessed by the Canadian Cardiovascular Society Scale (CCS) class, which ranges from grade I to IV. A higher CCS grade indicates a greater severity of angina.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1-Year after implantation
  Safety outcomes were defined as procedural final serious complications (perforation, abrupt closure, slow flow or no-reflow, unstable ventricular arrhythmias) and device failure (inability to cross coronary sinus, inability to expand; unplanned relocation of the device)
Change in potential aerobic capacity and endurance - The six minute walking test (6MWT) | 1-Year after implantation
  Change in subjects aerobic capacity and endurance will be assessed using The six minute walking test (6 MWT)- The longer the distance covered, the better the exercise tolerance
Reducing the severity of angina and it impact on quality of life, as shown by the Seattle Angina Questionnaire. | 1-Year after implantation
  Potential physical and quality of life limitations will be assessed using Seattle Angina Questionnaire-7 (SAQ-7). Summary score can best be understood by categorizing the scores into ranges: 0 to 24 represents poor health status, 25 to 49 as fair, 50 to 74 as good, and 75 to 100 as excellent.

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Department of Cardiology, The Copper Health Centre (MCZ), Lubin, Lower Silesian Voivodeship
  - Cardiac Department of Copper Health Center, Lubin, Lower Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wlodarczak S, Rola P, Jastrzebski A, Woitek F, Barycki M, Furtan L, Doroszko A, Wlodarczak A, Grygier M, Lesiak M. Coronary Sinus Reducer implantation in refractory angina: Short-term outcomes based on the Lower Silesia Sinus Reducer Registry (LSSRR). Kardiol Pol. 2023;81(5):508-511. doi: 10.33963/KP.a2023.0057. Epub 2023 Mar 5. No abstract available. PMID 36871301
- [Derived] Wlodarczak S, Rola P, Jastrzebski A, Barycki M, Furtan L, Wlodarczak P, Kulczycki JJ, Korda A, Turkiewicz K, Wlodarczak A, Lesiak M. Effectiveness of coronary sinus reducer implantation in routine clinical practice: 12-month outcomes. Pol Arch Intern Med. 2025 May 29;135(5):16986. doi: 10.20452/pamw.16986. Epub 2025 Apr 4. PMID 40192527